CLINICAL TRIAL: NCT06665386
Title: Prognostic Biomarkers for Selective Intra-Arterial Cooling Infusion Combined with Endovascular Thrombectomy in Acute Ischemic Stroke Based on Proteomics and Metabolomics.
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, MD.PhD, Capital Medical University
Other Study IDs: PBIA
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Hypothermia Treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Patients will receive best medical management (BMM) plus EVT according to the clinical guidelines.
- IA-SCI group: Patients will receive BMM and EVT combined with selective intra-arterial cold saline infusion.
  Interventions: Procedure: hypothermia

INTERVENTIONS:
Procedure: hypothermia — Patients who meet the inclusion criteria and do not meet the exclusion criteria will be randomly assigned to either the control group or the IA-SCI group. Control group patients will receive BMM and EVT. IA-SCI group patients will receive BMM and EVT, and additionally a selective intraarterial cooling infusion. The specific method is as follows:
  * Pre-recanalization: During the procedure, a micro-catheter used to deploy the stent retriever is threaded coaxially into the common femoral artery through the guide catheter. The microcatheter is advanced over a microguide wire, traveling up through the neck until it reaches beyond the clot. A 50 mL cold 0.9% saline (4℃) is infused into the ischemic territory at a rate of 10 mL/min via the microcatheter. This enables the cold solution to infuse into the ischemic territory prior to revascularization.
  * Post-recanalization: Following vessel recanalization, cold 0.9% saline (4 ℃) is reinfused into the vessel via the catheter at a rate of 22 mL
  Groups: IA-SCI group

SUMMARY:
Endovascular Thrombectomy has emerged as a pivotal treatment modality for acute ischemic stroke. However, despite successful thrombus removal, a substantial proportion of patients still experience poor outcomes. Selective intra-arterial cooling has shown promise in decelerating stroke progression and providing neuroprotection. This study aims to identify biomarkers associated with the combination of selective intra-arterial cooling infusion and endovascular thrombectomy in the treatment of ischemic stroke by integrating proteomics and metabolomics data. Our study is based on the multicenter RCT study "Safety and Efficacy of Selective Intra-Arterial Cooling Infusion Combined With EVT in Acute Ischemic Stroke." All samples were derived from this experiment. Our objective is to elucidate the molecular mechanisms underlying the prognostic impact of this combined therapeutic approach, providing insights to optimize stroke treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤80.
* Clinical signs consistent with acute ischemic stroke with large vessel occlusion in the anterior circulation (intracranial segment of the internal carotid artery, middle cerebral artery M1 segment) demonstrated with CTA/MRA/DSA.
* NIHSS score obtained prior to randomization ≥6 and ≤25.
* Modified Rankin Scale ≤ 1 prior to qualifying stroke.
* Arterial puncture performed within 24 hours from symptom onset or LKW.
* For the patients with symptom onset within 6 hours, the ASPECT score ≥6; for the patientswith onset within 6-24 hours, the therapy should meet the imaging criteria of DAWN or DEFUSE-3 trial.
* Patient/Legally Authorized Representative has signed the Informed Consent Form.

Exclusion Criteria:

* Baseline CT/MRI confirms the presence of multiple vascular territory acute strokes.
* Baseline CT/MRI confirms the presence of arterial dissection.
* Evidence of intracranial hemorrhage or hemorrhagic transformation before thrombectomy.
* Known allergies or intolerances to antiplatelet agents, anticoagulation drugs, iodinated contrast and/or anesthetics.
* Severe infection (e.g. sepsis) or multiple organ failure.
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR > 3. Patients on factor Xa inhibitor for 48 hours ago must have a normal APTT.
* Baseline platelet count <50 × 109/L.
* Blood glucose concentration<50 mg/dL (2.7mmol/L) or >400 mg/dL (22.2mmol/L).
* Refractory hypertension that is difficult to control by medication (Defined as persistent systolic blood pressure>185 mmHg or diastolic blood pressure>110mmHg).
* Previous NHYA>1.
* Untreated moderate or severe coronary artery stenosis, or previous coronary artery bypass surgery.
* Undergoing hemodialysis or peritoneal dialysis; known severe renal insufficiency with glomerular filtration rate <30 ml/min or serum creatinine >220 mmol/L (2.5mg/dl).
* Known intracranial aneurysm, and cerebral arteriovenous malformation.
* Malignant brain tumor or CNS infection.
* Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations (e.g., dementia or mental illness)
* Female who is pregnant or lactating at time of admission.
* Anticipated life expectancy <6 months.
* Current participation in another investigational drug or device study.
* For other reasons, the responsible clinicians believe that the patient is not suitable for continued treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood samples were collected from patients who underwent Endovascular Thrombectomy alone and those who received selective intra-arterial cooling infusion combined with Endovascular Thrombectomy. The supernatant was separated by centrifugation and stored in a -80°C refrigerator.
Sampling Method: Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 2024-10-2025-2
  Prognostic Biomarkers for Selective Intra-Arterial Cooling Infusion Combined with Endovascular Thrombectomy in Acute Ischemic Stroke Based on Proteomics and Metabolomics.
  Measure Description:
  By integrating proteomics and metabolomics data, researchers were able to identify common pathways and mechanisms through which selective intra-arterial cooling infusion combined with endovascular thrombectomy influences the prognosis of ischemic stroke.
  Time Frame:3 months

SECONDARY OUTCOMES:
Secondary Outcome | 2024-10-2025-2
  1. Quantitative changes of individual metabolites and proteins were calculated and graphed using the KEGG mapping tools.
  2. All of the omics data were used to compare proteins/enzymes with metabolic pathways.
  3. By integrating proteomics and metabolomics data, researchers were able to identify common pathways and mechanisms through which selective intra-arterial cooling infusion combined with endovascular thrombectomy influences the prognosis of ischemic stroke.
  Time Frame:3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dalian Municipal Central Hospital, Dalian, Liaoning, China